CLINICAL TRIAL: NCT01104649
Title: Efficacy of Riluzole in Hereditary Cerebellar Ataxia: a Randomized Double-blind Placebo-controlled Trial.
Brief Title: Efficacy of Riluzole in Hereditary Cerebellar Ataxia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Giovanni Ristori, MD, PhD, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FARM7KAJM7
Record Dates: First submitted 2010-04-07; First posted 2010-04-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Cerebellar Ataxia
Keywords: Spinocerebellar ataxia; Friedreich ataxia
MeSH Terms: conditions — Cerebellar Ataxia; Spinocerebellar Ataxias; Friedreich Ataxia | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Experimental): Riluzole 50 mg is administered orally every 12 hours for 12 months (a 2:1 ratio for SCA/FA in the stratified randomization procedure)
  Interventions: Drug: riluzole
- Placebo comparator (Placebo Comparator): Placebo is administered orally every 12 hours for 12 months (a 2:1 ratio for SCA/FA in the stratified randomization procedure)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: riluzole — Study drug will be orally dispensed in doses of 50 mg twice daily for 12 months.
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo comparator — Study drug will be orally dispensed in doses of 50 mg twice daily for 12 months.
  Other Names: Placebo
  Arms: Placebo comparator

SUMMARY:
The hereditary cerebellar ataxias include diverse neurodegenerative disorders. Hereditary ataxias can be divided into autosomal dominant ataxias (ADCAs), autosomal recessive ataxias (ARCAs), X-linked, and mitochondrial ataxias on the basis of mode of inheritance. The key feature in all these disorders is ataxia typically characterised by poor balance, hand incoordination, postural or kinetic tremor, dysarthria and dysphagia.

To date no treatment has been shown to slow progression of the disease and symptomatic therapies are limited to few options that are partially effective.

Purkinje cells project inhibitory signals to the deep cerebellar nuclei(DCN) which have a critical role in cerebellar function and motor performance. DCN neurons fire spontaneously in the absence of synaptic input from Purkinje neurons and modulation of the DCN response by Purkinje input is believed to be responsible for coordination of movement, while uncontrolled spontaneous firing of DCN neurons may underlay cerebellar ataxia. Recent studies have demonstrated that small-conductance calcium-activated potassium (SK) channels inhibitor are able to increase DCN firing rate. Since SK channels are critical regulators of DCN firing rate, SK openers such as the drug riluzole may reduce neuronal hyperexcitability and thereby be useful in the therapy of cerebellar ataxia.

On this base the investigators published a pilot study in patients with chronic cerebellar ataxia (Ristori et al., Neurology 2010) investigating safety and efficacy of riluzole or placebo administration for 8 weeks. The results demonstrated a significative improvement in International Cooperative Ataxia Rating Scale (ICARS) global score after four weeks and after 8 weeks in the riluzole arm.

The present protocol is aimed at verifying the safety and efficacy of riluzole administration for a longer period, in a larger sample size of patients, with more stringent diagnostic criteria (hereditary cerebellar ataxia), respect to the above pilot study. Sixty patients will be enrolled in a double-blind, placebo-controlled trial. By central randomisation, patients will take 50 mg of riluzole or placebo twice daily for 12 months. Treatment effects will be assessed by comparing the Scale for the Assessment and Rating of Ataxia (SARA) before treatment and during therapy at months 3 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically confirmed diagnosis of hereditary cerebellar ataxia

Exclusion Criteria:

* Concomitant experimental therapy for ataxia
* Serious systemic illnesses
* Pregnancy

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) | 12 months
  Improvement in ataxia

SECONDARY OUTCOMES:
Baropodometric parameters | 12 months
Quality of life | 12 months
  SF-36
Depression | 12 months
  Beck Scale

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Romano, MD, PhD, Principal Investigator — Center for Experimental Neurological Therapies (CENTERS), S. Andrea Hospital, II Faculty of Medicine, "Sapienza" University of Rome
Locations (1):
- Center for Experimental Neurological Therapies (CENTERS), S. Andrea Hospital, II Faculty of Medicine, "Sapienza" University of Rome, Rome, Italy

REFERENCES:
- [Background] Ristori G, Romano S, Visconti A, Cannoni S, Spadaro M, Frontali M, Pontieri FE, Vanacore N, Salvetti M. Riluzole in cerebellar ataxia: a randomized, double-blind, placebo-controlled pilot trial. Neurology. 2010 Mar 9;74(10):839-45. doi: 10.1212/WNL.0b013e3181d31e23. PMID 20211908
- [Derived] Romano S, Coarelli G, Marcotulli C, Leonardi L, Piccolo F, Spadaro M, Frontali M, Ferraldeschi M, Vulpiani MC, Ponzelli F, Salvetti M, Orzi F, Petrucci A, Vanacore N, Casali C, Ristori G. Riluzole in patients with hereditary cerebellar ataxia: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2015 Oct;14(10):985-91. doi: 10.1016/S1474-4422(15)00201-X. Epub 2015 Aug 25. PMID 26321318